CLINICAL TRIAL: NCT05693064
Title: The Impact of Chiropractic on Fatigue & the Autonomic Nervous System in Adults With Long COVID-19: a Waitlist-controlled, Single-blind, One-way Crossover, Pilot Trial
Brief Title: The Impact of Chiropractic on Long COVID-19
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding is needed before continuing
Sponsor: Life University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-0021
Record Dates: First submitted 2023-01-18; First posted 2023-01-20 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Waiting Lists; Manipulation, Chiropractic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wait-list followed by chiropractic (Experimental)
  Interventions: Other: wait-list; Procedure: chiropractic adjustments

INTERVENTIONS:
Other: wait-list — wait-list
Procedure: chiropractic adjustments — chiropractic adjustments

SUMMARY:
The purpose of this waitlist-controlled, single-blind, one-way crossover, pilot trial is to evaluate the potential effects of ~8 weeks of chiropractic care on patient-reported fatigue and the autonomic nervous system in adults with long COVID. This study will allow us to estimate the standard deviation of the primary endpoint in our population with which a formal power calculation for a future randomized, controlled trial can be performed.

DETAILED DESCRIPTION:
After providing informed consent, participants will be placed on an 8-week waitlist followed by 8 weeks of chiropractic care. In-person assessments will occur 5 times: Day 1, following 2-3 weeks on waitlist, following 8 weeks on waitlist, following 2-3 weeks of chiropractic care, and following 8 weeks of chiropractic care. Patient-reported outcomes will additionally be sent prior to the first in-person assessment (Day 0).

Assessments will include the following:

1. Seated resting recording
2. Sit-to-stand test
3. Patient-reported outcome surveys

Each assessment will consist of the following recordings:

1. Electroencephalography [EEG]
2. Impedance cardiography [ICG]
3. Electrocardiogram [ECG]

ELIGIBILITY:
Participants will be individuals between the age of 18 and 65 who have tested positive for a COVID-19 viral infection, or SARS-CoV-2 antibodies, not less than 120 days prior to their enrollment in the study. Participants may also qualify if they have been medically diagnosed with long-COVID by their medical provider, regardless of a positive test result. They must have a T score greater than or equal to 55 on the FACIT Fatigue survey. They must also present with at least 1 of the following symptoms that cannot be explained by an alternative diagnosis, with symptom onset or exacerbation after contraction of COVID-19.

* Body aches/joint pain
* Shortness of breath or difficulty breathing
* Persistent chest pain or pressure
* Recurrent fever, chills or night sweats
* Headache or dizziness
* Difficulty concentrating or focusing
* Memory problems
* Sleep problems
* Anxiety or depression
* Heart palpitations or tachycardia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
FACIT fatigue scale | Preliminary
  Patient Reported Outcome - The FACIT Fatigue Scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a 4-point Likert scale (4 = not at all fatigued to 0 = very much fatigued)
FACIT fatigue scale | Baseline (Day 1)
  Patient Reported Outcome - The FACIT Fatigue Scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a 4-point Likert scale (4 = not at all fatigued to 0 = very much fatigued)
FACIT fatigue scale | 2-3 weeks on wait-list
  Patient Reported Outcome - The FACIT Fatigue Scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a 4-point Likert scale (4 = not at all fatigued to 0 = very much fatigued)
FACIT fatigue scale | 8 weeks on wait-list
  Patient Reported Outcome - The FACIT Fatigue Scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a 4-point Likert scale (4 = not at all fatigued to 0 = very much fatigued)
FACIT fatigue scale | 2 - 3 weeks following start of intervention
  Patient Reported Outcome - The FACIT Fatigue Scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a 4-point Likert scale (4 = not at all fatigued to 0 = very much fatigued)
FACIT fatigue scale | Post intervention
  Patient Reported Outcome - The FACIT Fatigue Scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a 4-point Likert scale (4 = not at all fatigued to 0 = very much fatigued)

SECONDARY OUTCOMES:
EEG resting state broadband power | Baseline (Day 1)
  256-channel hydronet cap
EEG resting state broadband power | 2-3 weeks on wait-list
  256-channel hydronet cap
EEG resting state broadband power | 8 weeks on wait-list
  256-channel hydronet cap
EEG resting state broadband power | 2 - 3 weeks following start of intervention
  256-channel hydronet cap
EEG resting state broadband power | Post intervention
  256-channel hydronet cap
EEG resting state functional connectivity | Baseline (Day 1)
  256-channel hydronet cap
EEG resting state functional connectivity | 2-3 weeks on wait-list
  256-channel hydronet cap
EEG resting state functional connectivity | 8 weeks on wait-list
  256-channel hydronet cap
EEG resting state functional connectivity | 2-3 weeks following start of intervention
  256-channel hydronet cap
EEG resting state functional connectivity | Post intervention
  256-channel hydronet cap
ECG mean interbeat interval | Baseline (Day 1)
  3 sensors on torso
ECG mean interbeat interval | 2-3 weeks on wait-list
  3 sensors on torso
ECG mean interbeat interval | 8 weeks on wait-list
  3 sensors on torso
ECG mean interbeat interval | 2-3 weeks following start of intervention
  3 sensors on torso
ECG mean interbeat interval | Post intervention
  3 sensors on torso
ECG respiratory sinus arrhythmia (RSA) | Baseline (Day 1)
  3 sensors on torso
ECG respiratory sinus arrhythmia (RSA) | 2-3 weeks on wait-list
  3 sensors on torso
ECG respiratory sinus arrhythmia (RSA) | 8 weeks on wait-list
  3 sensors on torso
ECG respiratory sinus arrhythmia (RSA) | 2-3 weeks following start of intervention
  3 sensors on torso
ECG respiratory sinus arrhythmia (RSA) | Post intervention
  3 sensors on torso
Impedance cardiogram (ICG) pre-ejection period (PEP) | Baseline (Day 1)
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) pre-ejection period (PEP) | 2-3 weeks on wait-list
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) pre-ejection period (PEP) | 8 weeks on wait-list
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) pre-ejection period (PEP) | 2-3 weeks following start of intervention
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) pre-ejection period (PEP) | Post intervention
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) initial systolic time interval (ISTI) | Baseline (Day 1)
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) initial systolic time interval (ISTI) | 2-3 weeks on wait-list
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) initial systolic time interval (ISTI) | 8 weeks on wait-list
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) initial systolic time interval (ISTI) | 2-3 weeks following start of intervention
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) initial systolic time interval (ISTI) | Post intervention
  2 sensors on chest and 2 sensors on back
Patient-reported outcomes | Preliminary
  4 questionnaires - MFSI, IPAQ-S, PSS-4, C19-YRSm
Patient-reported outcomes | Baseline (Day 1)
  4 questionnaires - MFSI, IPAQ-S, PSS-4, C19-YRSm
Patient-reported outcomes | 2-3 weeks on wait-list
  4 questionnaires - MFSI, IPAQ-S, PSS-4, C19-YRSm
Patient-reported outcomes | 8 weeks on wait-list
  5 questionnaires - MFSI, IPAQ-S, PSS-4, C19-YRSm, GRC
Patient-reported outcomes | 2-3 weeks following start of intervention
  4 questionnaires - MFSI, IPAQ-S, PSS-4, C19-YRSm
Patient-reported outcomes | Post intervention
  5 questionnaires - MFSI, IPAQ-S, PSS-4, C19-YRSm, GRC

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Sullivan, DC, PhD, Study Director — Life Univeristy
Locations (1):
- Lydian Chiropractic LLC, Cambridge, Massachusetts, United States